CLINICAL TRIAL: NCT03761576
Title: The Role of Cognitive Function and Electroencephalography on Acute and Chronic Pain After Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Yi Feng, MD (Other)
Responsible Party: Sponsor-Investigator, Yi Feng, MD, director of department of anesthesiology and painmanagement, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Other Study IDs: 2018PHB191-02
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Acute Pain; Chronic Pain; Thoracic Surgery; Electroencephalography; Brain Mechanism
MeSH Terms: conditions — Acute Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The project will apply the methods of clinical observation experiment, (1) to collect the cognitive function data preoperatively and early postoperatively, as well as the pain score data at multiple time points pre- and postoperatively, and to observe the role of the degree of recovery of early postoperative cognitive function on acute pain and chronic pain after surgery. (2) to collect the resting-state electroencephalography (EEG) preoperatively, and to assess the role of EEG index system on the prediction of the degree of recovery of early postoperative cognitive function as well as the acute pain and chronic pain after surgery.

DETAILED DESCRIPTION:
Patients after surgery are liable to suffer from moderate to severe acute pain and refractory chronic pain, which would lead to serious somatic and psychological suffering. Its successful treatment is a great challenge for pain physicians. To date, the mechanism of pain chronification after surgery remains unclear. Further, it is still lack of efficient preventive and therapeutic measures for this chronic pain. The project will apply the methods of clinical observation and animal experiment, (1) to collect the cognitive function data preoperatively and early postoperatively, as well as the pain score data at multiple time points pre- and postoperatively, and to observe the role of the degree of recovery of early postoperative cognitive function on acute pain and chronic pain after thoracic surgery. (2) to collect the resting-state electroencephalography (EEG) preoperatively, and to assess the role of EEG index system on the prediction of the degree of recovery of early postoperative cognitive function as well as the acute pain and chronic pain after thoracic surgery. The project will be able to determine the relationships between the degree of recovery of early postoperative cognitive function, as well as preoperative resting-state EEG indices and postoperative acute pain and chronic pain, and clarify the neural mechanism of acute pain and chronic pain after surgery. The expected outcomes of this study can contribute to early identification of the patients who are liable to develop into acute pain and chronic pain after surgery, and give them reasonable intervention in time, and provide effective solutions for the acute pain and chronic pain after surgery.

ELIGIBILITY:
Inclusion Criteria:

* surgery were planned to be performed under general anesthesia
* Educational attainment beyond high school
* Require postoperative analgesia and sign the informed consent

Exclusion Criteria:

* with mental illness or a family history of mental illness
* Patients with cerebrovascular diseases or cerebrovascular accidents
* Previous head trauma history or craniotomy
* Using central analgesics, opioids addiction
* With a history of alcoholism
* do not understand the numerical rating scale(NRS) score and can not use patient-controlled analgesia(PCA）

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-21 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
acute pain | the third day of the surgery
  numerical rating scale(NRS)>3
chronic pain | the second month of the surgery
  numerical rating scale(NRS)>3

CONTACTS AND LOCATIONS:
Overall Officials: Yi Feng, MD, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang YQ, Li YR, Han Q, Gao F, Feng Y. Evaluation of dynamic brain function in patients with different degrees of chronic pain by EEG microstate analysis. BMC Anesthesiol. 2025 Oct 14;25(1):491. doi: 10.1186/s12871-025-03326-1. PMID 41087907
- [Derived] Han Q, Yue L, Gao F, Zhang L, Hu L, Feng Y. The Prediction of Acute Postoperative Pain Based on Neural Oscillations Measured before the Surgery. Neural Plast. 2021 Apr 9;2021:5543974. doi: 10.1155/2021/5543974. eCollection 2021. PMID 33897775